CLINICAL TRIAL: NCT01809015
Title: A Study Programme for the Evaluation of Oral Anticoagulation Therapy With Vitamin K Antagonists
Brief Title: Evaluation of Oral Anticoagulation With Vitamin K Antagonists - The thrombEVAL Study Programme
Acronym: thrombEVAL
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Ministry of Health, Rhineland-Palatinate, Germany (Unknown); Ministry of Economics, Rhineland-Palatinate, Germany (Unknown); German Federal Ministry of Education and Research (Other Government); Boehringer Ingelheim (Industry); Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry); Sanofi (Industry); IMO Institut GmbH (Unknown); PortaVita BV (Unknown); The German Heart Foundation (Other); Bayer (Industry)
Responsible Party: Principal Investigator, Philipp Wild, MD, MSc, Univ.-Prof. Dr. med. Philipp Wild, MSc, Johannes Gutenberg University Mainz
Other Study IDs: UMCM-2010EPI01
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Anticoagulant Antagonists, Vitamin K and Other Coagulants Causing Adverse Effects in Therapeutic Use; Atrial Fibrillation; Venous Thromboembolism
Keywords: Oral Anticoagulation; Regular Medical Care; Coagulation Service; Vitamin-K Antagonists; Quality of therapy; Atrial fibrillation; Venous thromboembolism; Bypass surgery; Prosthetic heart valve
MeSH Terms: conditions — Atrial Fibrillation; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cohort A: Regular medical care: Patients treated with vitamin K antagonists in regular medical care system
- Cohort B: Coagulation service: Patients with oral anticoagulation therapy in a telemedicine-based coagulation service

SUMMARY:
Since decades, oral anticoagulation (OAC) with vitamin K antagonists (VKA) is an established therapy for both prevention and treatment of thromboembolism in daily clinical routine. Increasing life-expectancy, the demographic change and novel oral anticoagulants lead to an increasing complexity of medical therapy. However, data on quality and management of VKA therapy with phenprocoumon in current medical care are limited. Our aim was to investigate the quality of OAC with VKA in current health care and to evaluate the potential for improvements.

The investigator-initiated thrombEVAL study program comprises two cohorts of patients treated with vitamin K antagonists for oral anticoagulation therapy in real-life settings: a multicentre cohort of patients in regular medical care and a multi-local, single centre cohort of patients in a telemedicine-based coagulation service. The study program is expected to enrol a total number of approximately 2,000 to 2,500 patients. Both cohorts build on a detailed clinical assessment of participants and anticoagulation therapy at study enrolment. Subsequently active and passive follow-up investigations are carried out to document and validate complications of the treatment. Primary short-term outcome is the distribution of time in therapeutic range; the primary long-term outcome comprises the composite of stroke, systemic embolism, myocardial infarction, major and clinically-relevant bleeding and death.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years of age at study inclusion
2. Written informed consent by patient or legal guardian, if appointed
3. Cohort A: Pretreatment with oral anticoagulation therapy with vitamin K antagonists (VKA) for at least 4 months in regular medical care including patients with self-management of oral anticoagulation therapy
4. Cohort B: Indication for oral anticoagulation therapy with VKA for at least 3 months (both drug-naive and -experienced patients) at enrolment including patients with self-management of oral anticoagulation therapy.

Exclusion Criteria

1. Contraindication to VKA treatment, e.g. pregnancy or known hypersensitivity
2. Participation in other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In cohort A, patients of regular medical care are enrolled in the area of Rhineland-Palatinate, Germany. Treatment and management of oral anticoagulation therapy with vitamin K antagonists is performed within primary (ambulatory) care system.
  In cohort B, patients are treated with oral anticoagulation in a specialized telemedicine-based coagulation service in the area of Rhinehesse, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 2318 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Time in therapeutic range | Assessment during Year 1 after study enrolment
  Time in therapeutic range for the International Normalized Ratio as measured by linear interpolation method
Hospitalisation | Assessment at year 1 and 2 after study enrolment
  Any Hospitalisation
Net clinical benefit | Assessment at year 1 and 2
  Composite of stroke, systemic embolism, pulmonary embolism, myocardial infarction, major and clinically relevant, non-major bleeding and death

CONTACTS AND LOCATIONS:
Overall Officials: Philipp S Wild, MD, MSc, Principal Investigator — University Medical Center of Johannes Gutenberg-University Mainz, Germany; Thomas F Munzel, MD, Principal Investigator — University Medical Center of Johannes Gutenberg-University Mainz, Germany
Locations (1):
- University Medical Center of the Johannes Gutenberg University Mainz, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Derived] Keller K, Prochaska JH, Coldewey M, Gobel S, Schmitt VH, Hahad O, Ullmann A, Nagler M, Lamparter H, Espinola-Klein C, Munzel T, Wild PS. Atherosclerosis and Its Impact on the Outcomes of Patients with Deep Venous Thrombosis. Life (Basel). 2022 May 14;12(5):734. doi: 10.3390/life12050734. PMID 35629401
- [Derived] Eggebrecht L, Ludolph P, Gobel S, Panova-Noeva M, Arnold N, Nagler M, Bickel C, Lauterbach M, Hardt R, Cate HT, Lackner KJ, Espinola-Klein C, Munzel T, Prochaska JH, Wild PS. Cost saving analysis of specialized, eHealth-based management of patients receiving oral anticoagulation therapy: Results from the thrombEVAL study. Sci Rep. 2021 Jan 28;11(1):2577. doi: 10.1038/s41598-021-82076-9. PMID 33510343
- [Derived] Michal M, Eggebrecht L, Gobel S, Panova-Noeva M, Nagler M, Arnold N, Lauterbach M, Bickel C, Wiltink J, Beutel ME, Munzel T, Wild PS, Prochaska JH. The relevance of depressive symptoms for the outcome of patients receiving vitamin K antagonists: results from the thrombEVAL cohort study. Eur Heart J Cardiovasc Pharmacother. 2021 Jul 23;7(4):271-279. doi: 10.1093/ehjcvp/pvz085. PMID 31922545
- [Derived] Prochaska JH, Gobel S, Nagler M, Knopfler T, Eggebrecht L, Lamparter H, Panova-Noeva M, Keller K, Coldewey M, Bickel C, Lauterbach M, Hardt R, Espinola-Klein C, Ten Cate H, Rostock T, Munzel T, Wild PS. Sustained atrial fibrillation increases the risk of anticoagulation-related bleeding in heart failure. Clin Res Cardiol. 2018 Dec;107(12):1170-1179. doi: 10.1007/s00392-018-1293-4. Epub 2018 Jun 9. PMID 29948286
- [Derived] Prochaska JH, Gobel S, Keller K, Coldewey M, Ullmann A, Lamparter H, Schulz A, Schinzel H, Bickel C, Lauterbach M, Michal M, Hardt R, Binder H, Espinola-Klein C, Lackner KJ, Ten Cate H, Munzel T, Wild PS. e-Health-based management of patients receiving oral anticoagulation therapy: results from the observational thrombEVAL study. J Thromb Haemost. 2017 Jul;15(7):1375-1385. doi: 10.1111/jth.13727. Epub 2017 Jun 6. PMID 28457013
- [Derived] Keller K, Prochaska JH, Coldewey M, Gobel S, Ullmann A, Junger C, Lamparter H, Ariza L, Bickel C, Lauterbach M, Konstantinides S, Rostock T, Munzel T, Wild PS. History of deep vein thrombosis is a discriminator for concomitant atrial fibrillation in pulmonary embolism. Thromb Res. 2015 Nov;136(5):899-906. doi: 10.1016/j.thromres.2015.08.024. Epub 2015 Sep 3. PMID 26376038
- [Derived] Prochaska JH, Gobel S, Keller K, Coldewey M, Ullmann A, Lamparter H, Junger C, Al-Bayati Z, Baer C, Walter U, Bickel C, ten Cate H, Munzel T, Wild PS. Quality of oral anticoagulation with phenprocoumon in regular medical care and its potential for improvement in a telemedicine-based coagulation service--results from the prospective, multi-center, observational cohort study thrombEVAL. BMC Med. 2015 Jan 23;13:14. doi: 10.1186/s12916-015-0268-9. PMID 25616558
- [Derived] Prochaska JH, Coldewey M, Gobel S, Keller K, Hendelmeier M, Konstantinides S, Munzel T, Wild PS; thrombEVAL Study Group. Evaluation of oral anticoagulation therapy: rationale and design of the thrombEVAL study programme. Eur J Prev Cardiol. 2015 May;22(5):622-8. doi: 10.1177/2047487314527852. Epub 2014 Mar 31. PMID 24685605
- See also: Study information homepage — http://www.thrombeval.de/